CLINICAL TRIAL: NCT05036863
Title: Feasibility Study of a Electronic Patient-Reported Outcome (ePRO) Monitoring for Patients With Multiple Myeloma and Development and Evaluation of Treatment-specific Item Lists
Brief Title: Feasibility Study of an ePRO Monitoring for Patients With Multiple Myeloma and Development of Item Lists
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: SymOn[2021]
Record Dates: First submitted 2021-06-24; First posted 2021-09-08 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-08

CONDITIONS: Multiple Myeloma
Keywords: Patient reported outcomes; Symptom monitoring; Follow-up; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with multiple myeloma
  Interventions: Behavioral: Weekly questionnaires

INTERVENTIONS:
Behavioral: Weekly questionnaires — Patients will complete weekly symptom monitoring PROMs. If a symptom exceeds the thresholds for clinical importance, a registered nurse will contact the patient, confirm the symptoms and coordinate the further clinical procedure in line with standard practice.

SUMMARY:
The trial is a feasibility study of a patient-reported outcome (PRO) monitoring for patients with multiple myeloma. Patients will report weekly PROs during treatment at our outpatient unit. The trial will describe the development of treatment-specific item lists to adequately capture relevant symptoms during therapy, evaluate the feasibility of the weekly symptom monitoring, and evaluate the healthcare professional usage of the system in clinical practice.

DETAILED DESCRIPTION:
The trial is a feasibility study of a patient-reported outcome (PRO) monitoring for patients with multiple myeloma. Patients will report weekly PROs during treatment at our outpatient unit. The trial will describe the development of treatment-specific item lists to adequately capture relevant symptoms during therapy, evaluate the feasibility of the weekly symptom monitoring, and evaluate the healthcare professional usage of the system in clinical practice.

The item lists will supplement an already established patient-reported outcome measure (PROM) implementation for the Austrian Myeloma Registry (AMR) at the Department of Hematology in Innsbruck. For the development of the treatment-specific item lists, a review of the literature for symptoms reported in clinical trials of the respective treatment regimens will be conducted. Then, a consensus panel of multiple stakeholders will discuss the symptoms and relevant issues for each treatment group. In an iterative process, the item lists will be developed to capture the most relevant and clinically important symptoms during active therapy to maximize clinical usage.

The observational part of the trial will then test the feasibility of the electronic symptom monitoring and the treatment-specific item lists. Patients will be recruited who are already participating in a routine care patient-reported outcome monitoring. They will be given access to the web-based patient portal and asked to complete weekly assessments using the treatment-specific item lists. In larger intervals (every 6 weeks), they will also be asked to complete a larger questionnaire battery using the EORTC QLQ-C30 and the treatment-specific module (EORTC QLQ-MY20). In the patient portal, patients will also be able to review their own results and receive feedback and self-management advice. Patients will also receive reminders to remind them to use the patient portal.

For healthcare professionals, the system will display the results of the PROMs and trigger alerts if patients reach thresholds for clinical importance. A clinical nurse will monitor the recently completed PROMs and contact patients who exceed the thresholds.

Patients will stay on the symptom monitoring as long as they receive active treatment. They may be excluded if they move to stationary care, depending on their health status or if they want to end the monitoring. The feasibility of the weekly monitoring and items lists will be evaluated and patient feedback to the patient portal and item lists will be recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed
* sufficient language proficiency in German
* no overt cognitive impairments
* reporting to use the internet at least once a month
* able to log into a website using an individualized username and password (tested when patients are introduced to the patient portal)
* patients are currently receiving active therapy for the treatment of their multiple myeloma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with multiple myeloma who meet the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Patient rated feasibility and adequacy of the item lists and symptom monitoring program | 6 weeks after inclusion of the patient or after the patient used the portal 3 times, whichever came first
  assessed via a questionnaire, after six weeks in the program or after using the portal 3 times (whichever occurs first); ratings are provided on a 1 to 4 scale ("not at all" to "very much", higher scores are better); the evaluation questionnaire was created for the study
Assessment completion rate | From the inclusion of the patient until the end of the study (ie, at maximum 12 months) or until the patient withdraws, whichever came first
  Calculated as the number of completed assessments divided by the number of expected assessments.

SECONDARY OUTCOMES:
Completeness of questionnaires | From the inclusion of the patient until the end of the study (ie, at maximum 12 months) or until the patient withdraws, whichever came first
  Number of missing items in the symptom item sets
Frequency of clinical alerts in the system | All alerts generated during the study period (ie, at maximum 12 months)
  The frequency of clinical alerts in the system (appropriateness of thresholds) and the interventions that were taken in response to the alerts will be investigated

CONTACTS AND LOCATIONS:
Locations (1):
- Hämatologische Ambulanz - Tirol Kliniken, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lehmann J, de Ligt KM, Tipelius S, Giesinger JM, Sztankay M, Voigt S, van de Poll-Franse LV, Rumpold G, Weger R, Willenbacher E, Willenbacher W, Holzner B. Adherence to Patient-Reported Symptom Monitoring and Subsequent Clinical Interventions for Patients With Multiple Myeloma in Outpatient Care: Longitudinal Observational Study. J Med Internet Res. 2023 Aug 22;25:e46017. doi: 10.2196/46017. PMID 37606979